CLINICAL TRIAL: NCT04817904
Title: Evaluation of the Effect of Rosuvastatin on Cisplatin-induced Nephrotoxicity and Ototoxicity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: German University in Cairo (Other)
Responsible Party: Principal Investigator, Aya Tarek Moustafa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S-4-2020
Record Dates: First submitted 2021-03-21; First posted 2021-03-26 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cisplatin Adverse Reaction
Keywords: cisplatin; rosuvastatin; nephrotoxicity; ototoxicity
MeSH Terms: conditions — Ototoxicity | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Statin-Treated (Experimental): This arm will be receiving:
  * Cisplatin along with conventional nephroprotective interventions (IV hydration with 3 liters with electrolyte replacement administered on the same day of cisplatin)
  * Rosuvastatin 10 mg/day
  Interventions: Drug: Rosuvastatin 10mg
- Statin-Free (No Intervention): This arm will be receiving:
  -Cisplatin along with conventional nephroprotective interventions only (IV hydration with 3 liters with electrolyte replacement administered on the same day of cisplatin)

INTERVENTIONS:
Drug: Rosuvastatin 10mg — The statin-treated arm will receive Rosuvastatin tablets 10 mg/day starting from the point of cisplatin initiation through the entire duration of therapy
  Arms: Statin-Treated

SUMMARY:
Cisplatin is an effective anti-cancer drug for the treatment of many solid tumors in humans. Although the clinical response to cisplatin chemotherapy is encouraging, the nephrotoxicity and ototoxicity of the drug makes it difficult to continue its administration in many cases.

Cisplatin nephrotoxicity occurs through several mechanisms, mainly through the transport and accumulation of cisplatin into renal epithelial cells, injury to nuclear and mitochondrial DNA, activation of multiple cell death pathways and initiation of inflammatory response. Accordingly, several experimental strategies were developed to prevent this toxicity. For example, drugs that reduced renal cisplatin accumulation such as organic cation transporter 2 (OCT2) and copper transporter (Ctr1) inhibitors, antioxidants, antiapoptotic and anti-inflammatory agents were investigated. However, many of these drugs interfered with the cytotoxic effects of cisplatin.

Statins are agents used for reducing plasma cholesterol through the inhibition of the enzyme 3- hydroxy-3- methylglutaryl coenzyme A (HMG-CoA) reductase. In addition, statins are also proven to have pleiotropic, non-lipid dependent effects. These effects include anti-inflammatory actions and reduction of oxidative stress. Based on animal studies performed, statins have been shown to reduce the nephrotoxic effects of cisplatin in rats. In addition, ongoing clinical trials are aiming to investigate the role of statins in the protection against the ototoxicity of cisplatin as well. Our aim is to assess the protective effect of statins on cisplatin-induced nephrotoxicity and ototoxicity in humans.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven lung and breast cancer patients indicated for cisplatin (4-6 cycles)
* Normal baseline serum creatinine levels
* Normal baseline audiometry
* Age between 18-70 years

Exclusion Criteria:

* Patients with more than one type of cancer
* Patients with prior chemotherapy treatment
* Treatment with statins within 12 months before assignment
* Treatment with fibrates within 4 weeks before assignment
* Pregnancy and Lactation
* Abnormal liver function tests or blood count

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of cisplatin-induced nephrotoxicity | 4 months
  Increase in serum creatinine by ≥0.3 mg/dL or 1.5-2 fold increase from baseline

SECONDARY OUTCOMES:
Difference in biological research markers between both arms | 4 months
  Measurement of total antioxidant capacity and malondialdehyde levels
Difference in sensory-neural hearing impairment in both arms | 4 months
  Audiometry assessment
Incidence of electrolyte imbalance in both arms | 4 months
  Reduction in magnesium level ˂1.8 mg/dL and potassium level ˂3.5 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Solayman, PhD, Study Chair — German University in Cairo; Loay Kassem, PhD, Principal Investigator — Cairo University; Dalia S Elhelw, PhD, Principal Investigator — German University in Cairo; Aya T Moustafa, BSc, Principal Investigator — German University in Cairo
Locations (1):
- Kasr El-Aini Center of Radiation Oncology and Nuclear Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] An Y, Xin H, Yan W, Zhou X. Amelioration of cisplatin-induced nephrotoxicity by pravastatin in mice. Exp Toxicol Pathol. 2011 Mar;63(3):215-9. doi: 10.1016/j.etp.2009.12.002. Epub 2010 Jan 8. PMID 20060696
- [Background] Fujieda M, Morita T, Naruse K, Hayashi Y, Ishihara M, Yokoyama T, Toma T, Ohta K, Wakiguchi H. Effect of pravastatin on cisplatin-induced nephrotoxicity in rats. Hum Exp Toxicol. 2011 Jul;30(7):603-15. doi: 10.1177/0960327110376551. Epub 2010 Jul 22. PMID 20650967
- [Background] Seckl MJ, Ottensmeier CH, Cullen M, Schmid P, Ngai Y, Muthukumar D, Thompson J, Harden S, Middleton G, Fife KM, Crosse B, Taylor P, Nash S, Hackshaw A. Multicenter, Phase III, Randomized, Double-Blind, Placebo-Controlled Trial of Pravastatin Added to First-Line Standard Chemotherapy in Small-Cell Lung Cancer (LUNGSTAR). J Clin Oncol. 2017 May 10;35(14):1506-1514. doi: 10.1200/JCO.2016.69.7391. Epub 2017 Feb 27. PMID 28240967
- [Background] Pabla N, Dong Z. Cisplatin nephrotoxicity: mechanisms and renoprotective strategies. Kidney Int. 2008 May;73(9):994-1007. doi: 10.1038/sj.ki.5002786. Epub 2008 Feb 13. PMID 18272962